CLINICAL TRIAL: NCT04503395
Title: Physician Initiated Trial Investigating ESAR (EVAR Plus Heli-FX EndoAnchors) and FEVAR for the Treatment of Aortic Aneurysms With Short Infrarenal Aortic Neck
Brief Title: ShOrt neCK AAA RAndomized Trial - ESAR and FEVAR: SOCRATES
Acronym: SOCRATES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FCRE (Foundation for Cardiovascular Research and Education) (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Marc Bosiers, MD, Principal Investigator, FCRE (Foundation for Cardiovascular Research and Education)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCRE-191125
Record Dates: First submitted 2020-07-22; First posted 2020-08-07 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Aortic Aneurysm, Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Intervention Model Description: comparision of two different procedure to repair abdominal aortic aneurysms with short necks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ESAR (Experimental): Endovascular Aneurysm Repair + Heli-FX EndoAnchors
  Interventions: Device: ESAR treatment: Endograft + Heli-FX Endoanchor
- FEVAR (Active Comparator): Fenestrated EndoVascular Aneurysm Repair
  Interventions: Device: FEVAR treatment : Fenestrated endograft

INTERVENTIONS:
Device: ESAR treatment: Endograft + Heli-FX Endoanchor — ESAR treatment: Endurant II or Endurant IIs endograft + Heli-FX Endoanchor
  Arms: ESAR
Device: FEVAR treatment : Fenestrated endograft — Cook Zenith Fenestrated Graft or the Terumo Fenestrated Anaconda Graft
  Arms: FEVAR

SUMMARY:
The aim of this randomized study is to compare the safety and performance of EndoVascular Aneurysm Repair with ESAR using Endurant + Heli-FX™ EndoAnchor™ system and FEVAR using customizable grafts from Cook (Zenith Fenestrated Graft) and Terumo (Fenestrated Anaconda Graft) for the treatment of aortic aneurysms with short aortic neck (4 to 15mm).

ELIGIBILITY:
Inclusion Criteria:

* Subject is >18 years old
* Subject is scheduled for primary treatment of the abdominal aortic aneurysm with a non-aneurysmal infrarenal aortic sealing zone proximal to the aneurysm that is sufficiently healthy for a proximal neck length that is at least 4mm and not more than15 mm and has a circumferential minimum sealing zone length of 8 mm
* Subject is not a candidate for safe, effective and durable standard EVAR due to challenging anatomical criteria as confirmed by the Core Lab screening
* Subject is able and willing to comply with the protocol and to adhere to the follow-up requirements.
* Subject has provided written informed consent

CT Angiographic Inclusion Criteria

* Subject meets the other anatomical requirements according to the locally applicable Endurant II/IIs stent graft system, Heli-FX EndoAnchor system, Terumo Fenestrated Anaconda (available in EU only) and/or Cook Zenith Fenestrated Graft Instructions for Use
* Proximal neck length of the aorta within 4-15mm and a minimum circumferential sealing zone of 8mm
* Aortic neck diameter from 19 to 31mm
* Infrarenal neck angulation ≤45°

Exclusion Criteria:

* Subject is participating in a concurrent study which may confound study results
* Subject has a life expectancy <2 year
* Subject is female of childbearing potential in whom pregnancy cannot be excluded
* Subject with eGFR <30 mL/min/m2 (KDOQI classification - exclude class IV and above) and or on dialysis
* Subject with a MI or CVA within 3 months prior to index procedure
* Subject with known Connective Tissue Disease
* Subject has a known hypersensitivity or contraindication to anticoagulants, antiplatelets, or contrast media, which is not amenable to post-treatment
* Subject who has undergone prior endovascular or open surgical treatment for abdominal aortic aneurysm
* Subject requires emergent aneurysm treatment, for example, trauma or rupture
* Subject has a known hypersensitivity or allergies to study device implant material
* Subject has an aneurysm that is:

  * Suprarenal, pararenal, or thoracoabdominal
  * Mycotic
  * Inflammatory
  * Pseudoaneurysm
* Subject is presenting with thrombus or calcification of the proximal aneurysm neck: circumferential >50%
* Pre-op stenosis of the renal arteries > 50%
* Subject has active infection or history of COVID-19. History of COVID-19 is defined as availability of positive COVID-19 test with sequelae or hospitalization for treatment of COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness Endpoint - Technical Success | through 12 months post-procedure
  Composite of technical success at index procedure, and freedom from type IA or type III endoleak, freedom from aneurysm related mortality (ARM), and freedom from secondary reinterventions through 12 months post index procedure.
Safety Endpoint - Freedom from Major Adverse Events | through 30 days post-procedure
  Freedom from MAE through 30 days post index procedure. MAE defined as: All-Cause-Mortality, Bowel Ischemia, Myocardial Infraction, Procedural Blood Loss > 1000cc, Access related complications, permanent paraplegia and paraparesis at 30 days, disabling stroke, respiratory failure, or renal complications

SECONDARY OUTCOMES:
Total contrast volume (ml) at index procedure | at index procedure
  Total contrast volume (mL) at index procedure
Total fluoroscopy time (minutes) at index procedure | at index procedure
  Total fluoroscopy time (minutes) at index procedure
Duration (minutes) of index procedure | at index procedure
  3. Duration (minutes) of index procedure (time between initial skin access to final closure of the last artery access site)
Adequate penetration of EndoAnchor implants as assessed by the Core Lab | at index procedure
  Adequate penetration of EndoAnchor implants as assessed by the Core Lab
Clinical success | through 30 days post-procedure
  7. Clinical success defined as technical success + freedom from intra-operative death and freedom from type IA/III endoleak in the first post-op image within 30 days.
Visceral artery patency or occlusion at 1, 12, 24 and 36 months follow-up | through 1,12,24 and 36-months post-op
  Visceral artery patency or occlusion at 1, 12, 24 and 36 months follow-up
Freedom from type Ia and III endoleaks at 1, 12, 24 and 36 months follow-up | through 1,12,24 and 36-months post-op
  Freedom from type Ia and III endoleaks at 1, 12, 24 and 36 months follow-up
Freedom from aneurysm related secondary reinterventions at 1, 12, 24 and 36 months follow-up | through 1,12,24 and 36-months post-op
  Freedom from aneurysm related secondary reinterventions at 1, 12, 24 and 36 months follow-up
Freedom from aneurysm related mortality at 1, 12, 24 and 36 months follow-up | through 1,12,24 and 36-months post-op
  Freedom from aneurysm related mortality at 1, 12, 24 and 36 months follow-up
Freedom from stent graft migration (>10mm change from 1-month follow-up imaging) at 12, 24 and 36 months follow-up | through 12,24 and 36-months post-op
  Freedom from stent graft migration (>10mm change from 1-month follow-up imaging) at 12, 24 and 36 months follow-up
Sac dynamics (>5mm change from 1-month follow-up imaging): increase, stable, decrease at 12, 24, and 36 months follow-up | through 12,24 and 36-months post-op
  Sac dynamics (>5mm change from 1-month follow-up imaging): increase, stable, decrease at 12, 24, and 36 months follow-up
Freedom from conversion to open repair at 1, 12, 24 and 36 months follow-up | through 1,12,24 and 36-months post-op
  Freedom from conversion to open repair at 1, 12, 24 and 36 months follow-up
Freedom from AAA rupture at 1, 12, 24 and 36 months follow-up | through 1,12,24 and 36-months post-op
  Freedom from AAA rupture at 1, 12, 24 and 36 months follow-up
Overall SCI rate, include transient events at 1 and 12 months follow-up | through 1 and 12 months post-op
  Overall SCI rate, include transient events at 1 and 12 months follow-up
Freedom from aortic neck-related secondary interventions | at 1-, 12-, 24- and 36-months follow-up
  reinterventions for Type IAa endoleak, migration of the proximal stent graft, and progression of disease in the infrarenal aortic neck; progression of disease is defined as enlargement of the infrarenal aortic neck compared to the first postprocedural CT scan, as measured by either diameter, surface and/or volume.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Torsello, Prof. Dr., Principal Investigator — Vascupedia; Brant Ullery, MD, MBA, Principal Investigator — Medical Director, Vascular Surgery Providence Heart and Vascular Institute
Locations (32):
- United States (10):
  - UCSD Medical Center Hillcrest, La Jolla, California
  - Stanford University, Stanford, California
  - University of Florida, Gainesville, Florida
  - Corewell Health (Spectrum), Grand Rapids, Michigan
  - Mount Sinai Hospital, New York, New York
  - Atrium Health Carolinas Medical Center, Charlotte, North Carolina
  - Oklahoma Heart, Tulsa, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Hospital Ottakring, Institute for Vascular Surgery, Vienna, Austria
- Belgium (2):
  - CRC thoracic Vascular Surgery, ZOL Genk, Genk
  - Universitair Ziekenhuis Gent, Thoracale en vasculaire heelkunde, Ghent
- France (4):
  - Amrois Paré Hospital (APHP), Boulogne
  - Service de Chirurgie Vasculaire et Endovasculaire CHU Gabriel-Montpied 58 rue Montalembert, Clermont-Ferrand
  - Hospices Civils de lyon - Hôpital Edouard Herriot, Lyon
  - Centre Hospitalier Universitaire de Rennes, Rennes
- Germany (3):
  - University Hospital RWTH Aachen, Aachen
  - University Hospital Leipzig, Leipzig
  - Martin Austermann, Münster
- Italy (5):
  - University of Bologna, IRCCS S. Orsola Hospital,, Bologna
  - Az. Ospedaliera San Martino, Genova, Genova
  - IRCCS Ospedale San Raffaele, Chirurgia Vascolare, Milan
  - Vascular Endovascular Surgery University of Perugia;, Perugia
  - Az.Osped.Univers.S.Giovanni, Turin, Turin
- Netherlands (2):
  - VUMC Amsterdam, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
- National Institute of Cardiology Warzwa, Warsaw, Poland
- Spain (3):
  - Hospital Ramon Y Cajal, Madrid
  - Hospital Universitario Donostia, San Sebastián
  - HOSPITAL CLINICO UNIVERSITARIO Valladolid, Valladolid
- Inselspital Bern, Universitätsklinik für Gefässchirurgie, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No